CLINICAL TRIAL: NCT01922128
Title: A Phase 1 Randomized, Double-masked, Vehicle-controlled, Dose Escalation Study of the Ocular Safety and Tolerability of MC-1101 in Medically Stable Individuals
Brief Title: Safety Study of a Topical Treatment for Dry Age Related Macular Degeneration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MacuCLEAR, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MC-1101-002
Record Dates: First submitted 2013-08-07; First posted 2013-08-14 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-04

CONDITIONS: Nonexudative Age-related Macular Degeneration
Keywords: Non-exudative, dry AMD

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Drug, MC-1101 (Active Comparator): One eye drop of Active comparator, 0.5% MC-1101, 2 times per day, 28 days; followed by one drop of 1% MC-1101, 2 times per day, 28 days.
  Interventions: Drug: MC-1101, Placebo
- Placebo (Placebo Comparator): One eye drop of Placebo comparator to MC-1101. Placebo contains all components of MC-1101 except for the active ingredient.
  Interventions: Drug: MC-1101, Placebo

INTERVENTIONS:
Drug: MC-1101, Placebo — One drop 0.5%; MC-1101; One drop 1.0% MC-1101, One drop Placebo

SUMMARY:
Study to evaluate the safety and tolerability of MC-1101, a potential topical treatment for non-edxudative age Related Macular Degeneration (AMD) in medically stable individuals.

DETAILED DESCRIPTION:
MC-1101 is a topical version of a previously approved anti-hypertensive drug that is intended to increase choroidal blood flow.

* A reduction of choroidal blood flow has been identified in patients with AMD
* This study will evaluate 0.5% and 1.0% potencies of MC-1101 delivered 2X per day.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects ≥ 50 and ≤ 85 years of age.
2. Women must be post-menopausal or surgically sterilized for 1 year or longer.
3. Best corrected distance visual acuity of 1.0 logMAR of better in each eye (20/200 Snellen equivalent).
4. Able and willing to sign informed consent and HIPAA authorization, follow study instructions and complete all study visits. A study visit may require several exams during the course of the day.
5. Able and willing to discontinue the use of all ocular medication(s) except for artificial tears at least one week prior to receiving the study treatment and for the entire course of the study.
6. General good health, as evaluated by the investigator, based on the medical history provided by the subject and any adjunctive testing carried out at the investigator's discretion.

Exclusion Criteria:

Ophthalmic:

1. Previous intravitreal injections of anti-VEGF therapies in either eye.
2. History of diabetes and or diabetic retinopathy > 10 years.
3. Ocular of laser surgery in either eye within 3 months of Visit 1.
4. Ocular injection in either eye of any medication within 3 months of Visit 1.
5. History of incisional glaucoma surgery in either eye.
6. Corneal, cataract or media opacification in either eye which limits an adequate view of the fundus in the opinion of the investigator.
7. Contraindications to pupil dilation in either eye.
8. Any ocular disease that requires ongoing treatment with topical ocular agents in either eye during the study. Patients using intermittent ocular medications must stop these medications for one week prior to Visit 2. Use of artificial tears 3 times daily or less for mild dry eye disease is allowed, but must not occur within ± 15 minutes from dosing of the investigational product).
9. Corneal disease, corneal irregularity or scarring that in the opinion of the investigator would make it difficult to accurately measure intraocular pressure (IOP) or visualize intraocular anatomy in either eye.
10. Presence of a Hudson-Stahli line in the corneal epithelium in either eye.

General/Systemic:

1. Female subjects who are menstruating.
2. Prior participation (participation is defined as being randomized to an investigational product) in any other study in the last 30 days.
3. Subjects unable to administer or have a caretaker administer the study eye drops.
4. Subjects who are unable to follow instructions or are unwilling and considered physically unable to return for all study visits for the duration of the study.
5. Clinically significant systemic disease that in the opinion of the investigator would interfere with the subject's ability to comply with the study requirements and or interpretation of the study results.
6. Clinically significant abnormal results of laboratory tests, available to the investigator, which in the investigator's judgment would prohibit the subject from safe participation in this trial.
7. Current or past use (more than 30 days) of chloroquine, hydroxychloroquine, chlorpromazine, thioridazine, quinine sulfate, clofazamine, cisplatin, carmustine, or deferoxamine.
8. Uncontrolled blood pressure with systolic value ≥ 170 and diastolic ≥ 100 mmHg. Repeated measurements are allowed if in the investigator's opinion the time interval between recent antihypertensive medication dosing and blood pressure measurements was insufficient to provide for efficacious hypertension reduction.
9. Subjects likely to undergo changes in systemic medications. All medications taken on a chronic basis must be stable for 30 days prior to Visit 2. Medications for an acute illness used within 30 days of Visit 1 must be discontinued prior randomization.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-09; Primary Completion 2013-11 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
No significant ocular or systemic adverse events in any of the 20 study subjects | 56 total days
  Assess the safety and tolerability of MC-1101 by evaluating the local ocular and systemic safety of MC-1101 0.5 % and 1 % in subjects in a dose escalation manner over 8 weeks of daily ocular exposure.

CONTACTS AND LOCATIONS:
Overall Officials: Ken Sall, MD, Principal Investigator — Sall Eye Center
Locations (1):
- Sall Eye Center, Artesia, California, United States